CLINICAL TRIAL: NCT04177238
Title: Effects of Oral Fruit Concentrate Supplementation on Cardiometabolic Parameters.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Lancashire (Other)
Responsible Party: Principal Investigator, Jonathan Sinclair, Principal Investigator - Professor of Sport, Exercise & Nutritional Sciences, University of Central Lancashire
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Cherry/ blueberry concentrate
Record Dates: First submitted 2019-11-21; First posted 2019-11-26 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — blueberry extract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Identical in taste and colour to the supplement juice, but with no anthocyanin content
  Interventions: Dietary Supplement: Fruit concentrate - either cherry or blueberry
- Cherry juice (Experimental): 30 mL of tart juice concentrate, which will be diluted with 100 mL of water - taken twice per day,
  Interventions: Dietary Supplement: Fruit concentrate - either cherry or blueberry
- Blueberry (Experimental): 30 mL of tart juice concentrate, which will be diluted with 100 mL of water - taken twice per day,
  Interventions: Dietary Supplement: Fruit concentrate - either cherry or blueberry

INTERVENTIONS:
Dietary Supplement: Fruit concentrate - either cherry or blueberry — Fruit (cherry or blueberry concentrate) supplement from a company named Active-Edge (https://active-edge.co.uk/).

SUMMARY:
Cardiovascular disease, type 2 diabetes mellitus and associated diseases combined are the leading health burden and cause of mortality worldwide; therefore, the necessity for an intervention is paramount. Dietary interventions to improve cardiometabolic health are highly sought after as they possess less risk than pharmacological drugs. Anthocyanins, found in high quantities in both tart cherries and blueberries are powerful antioxidants, that are potentially capable of improving cardiometabolic dysfunction. However, to date, no research has explored the cardiometabolic responses to tart cherry and blueberry supplementation.

Therefore, the primary purpose of the proposed investigation is to test the ability of oral tart cherry and blueberry supplementation to improve cardiometabolic parameters in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* 18 years of age and above
* Non-smoker
* BMI < 30
* Able to give informed consent

Exclusion Criteria:

* Pregnancy
* Diabetes or any other metabolic/ uncontrolled hypertensive conditions
* Food allergies to cherries or blueberries
* Habitual consumption of blueberries/ cherries and/or blueberry/ cherry products
* Not regularly taking medication or antioxidant supplements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2022-02-05 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Baseline
  Systolic and diastolic blood pressure - measured using a digital blood pressure monitor
% bodyfat | Baseline
  Participants percentage composition of fat - measured using bio-electrical impedance
% bodyfat | 20 days
  Participants percentage composition of fat - measured using bio-electrical impedance
Waist to hip ratio | Baseline
  Ratio of waist to hip circumference - measured using anthropocentric tape
Waist to hip ratio | 20 days
  Ratio of waist to hip circumference - measured using anthropocentric tape
Resting metabolic rate | Baseline
  Estimated daily calorie usage (Kcal) at rest - obtained using a metabolic cart through indirect calorimetry.
Resting metabolic rate | 20 days
  Estimated daily calorie usage (Kcal) at rest - obtained using a metabolic cart through indirect calorimetry.
Resting utilization of carbohydrates | Baseline
  % contribution of carbohydrate to daily calories - at rest - obtained using a metabolic cart through indirect calorimetry.
Resting utilization of carbohydrates | 20 days
  % contribution of carbohydrate to daily calories - at rest - obtained using a metabolic cart through indirect calorimetry.
Resting utilization of fats | Baseline
  % contribution of fats to daily calories - at rest - obtained using a metabolic cart through indirect calorimetry.
Resting utilization of fats | 20 days
  % contribution of fats to daily calories - at rest - obtained using a metabolic cart through indirect calorimetry.
Low-moderate intensity activity calories expended | Baseline
  Estimated calorie usage (Kcal) during low-moderate intensity walking exercise - obtained using a metabolic cart through indirect calorimetry.
Low-moderate intensity activity calories expended | 20 days
  Estimated calorie usage (Kcal) during low-moderate intensity walking exercise - obtained using a metabolic cart through indirect calorimetry.
Low-moderate intensity activity utilization of fats | Baseline
  % contribution of fats to calorie expenditure - during low-moderate intensity walking exercise - obtained using a metabolic cart through indirect calorimetry.
Low-moderate intensity activity utilization of fats | 20 days
  % contribution of fats to calorie expenditure - during low-moderate intensity walking exercise - obtained using a metabolic cart through indirect calorimetry.
Low-moderate intensity activity utilization of carbohydrates | Baseline
  % contribution of carbohydrates to calorie expenditure - during low intensity walking exercise - obtained using a metabolic cart through indirect calorimetry.
Low-moderate intensity activity utilization of carbohydrates | 20 days
  % contribution of carbohydrates to calorie expenditure - during low intensity walking exercise - obtained using a metabolic cart through indirect calorimetry.
Blood glucose | Baseline
  Capillary blood glucose - mmol/L
Blood glucose | 20 days
  Capillary blood glucose - mmol/L
Blood triglycerides | Baseline
  Capillary blood triglycerides - mmol/L
Blood triglycerides | 20 days
  Capillary blood triglycerides - mmol/L
Blood cholesterol (Total, HDL & LDL) | Baseline
  Capillary blood cholesterol - mmol/L
Blood cholesterol (Total, HDL & LDL) | 20 days
  Capillary blood cholesterol - mmol/L
Blood haemoglobin | Baseline
  Capillary blood haemoglobin - g/L
Blood haemoglobin | 20 days
  Capillary blood haemoglobin - g/L
Coop-Wonka chart | Baseline
  Psychological wellbeing - The Coop-Wonka chart is a six item questionnaire with a 1-5 scoring system for each thus the chart has a maximum score of 30 which indicates the lowest possible psychological Wellbeing.
Coop-Wonka chart | 20 days
  Psychological wellbeing - The Coop-Wonka chart is a six item questionnaire with a 1-5 scoring system for each thus the chart has a maximum score of 30 which indicates the lowest possible psychological Wellbeing.
Beck Depression Inventory | Baseline
  Psychological wellbeing - the Beck Depression Inventory is a 21 questionnaire with questions that range in scoring from 0-3, thus the maximum score is 63 which is the highest depression score possible.
Beck Depression Inventory | 20 days
  Psychological wellbeing - the Beck Depression Inventory is a 21 questionnaire with questions that range in scoring from 0-3, thus the maximum score is 63 which is the highest depression score possible.
State Trait Anxiety Inventory | Baseline
  Psychological wellbeing - the state trait anxiety inventory is a 40 item questionnaire with each question having a 1-4 score system, thus the maximum score is 80 which indicates the highest level of anxiety.
State Trait Anxiety Inventory | 20 days
  Psychological wellbeing - the state trait anxiety inventory is a 40 item questionnaire with each question having a 1-4 score system, thus the maximum score is 80 which indicates the highest level of anxiety.
Insomnia Severity Index | Baseline
  Sleep quality - The Insomnia Severity Index is a brief instrument designed to assess the severity of both nighttime and daytime components of insomnia. The Insomnia Severity Index is a 7-item self-report questionnaire yielding a total score ranging from 0 to 28.
Insomnia Severity Index | 20 days
  Sleep quality - The Insomnia Severity Index is a brief instrument designed to assess the severity of both nighttime and daytime components of insomnia. The Insomnia Severity Index is a 7-item self-report questionnaire yielding a total score ranging from 0 to 28.
Pittsburgh Sleep Quality Index | Baseline
  Sleep quality - The Pittsburgh Sleep Quality index, is a questionnaire that consists of 19 self-rated questions, grouped into 7 components. Each component is scored separately, weighted equally on a 0 - 3 scale and the scores of the 7 components are then added to give a global score, which has a range of 0 - 21 with higher scores indicating worse sleep quality.
Pittsburgh Sleep Quality Index | 20 days
  Sleep quality - The Pittsburgh Sleep Quality index, is a questionnaire that consists of 19 self-rated questions, grouped into 7 components. Each component is scored separately, weighted equally on a 0 - 3 scale and the scores of the 7 components are then added to give a global score, which has a range of 0 - 21 with higher scores indicating worse sleep quality.
Epworth Sleepiness Scale | Baseline
  Sleep quality - The Epworth Sleepiness Scale is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3) with a maximum score of 24.
Epworth Sleepiness Scale | 20 days
  Sleep quality - The Epworth Sleepiness Scale is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3) with a maximum score of 24.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Lancashire, Preston, Lancashire, United Kingdom

REFERENCES:
- [Derived] Sinclair J, Shadwell G, Dillon S, Allan R, Butters B, Bottoms L. Effects of Montmorency Tart Cherry and Blueberry Juice on Cardiometabolic Outcomes in Healthy Individuals: Protocol for a 3-Arm Placebo Randomized Controlled Trial. Int J Environ Res Public Health. 2021 Sep 16;18(18):9759. doi: 10.3390/ijerph18189759. PMID 34574679